CLINICAL TRIAL: NCT00260741
Title: Cannabis for Spasticity in Multiple Sclerosis: A Placebo-Controlled Study
Brief Title: Cannabis for Spasticity in Multiple Sclerosis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Discontinued due to non-enrollment.
Sponsor: Center for Medicinal Cannabis Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C00-DA-112; 200311404-4
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2007-04

CONDITIONS: Multiple Sclerosis
Keywords: cannabis; marijuana; Multiple Sclerosis; Spasticity
MeSH Terms: conditions — Multiple Sclerosis; Marijuana Abuse; Muscle Spasticity

INTERVENTIONS:
Drug: Smoked Cannabis

SUMMARY:
The purpose of this study is to learn if the use of inhaled cannabis (marijuana) and oral cannabinoid (dronabinol, Marinol or THC, which is an active ingredient of marijuana) is safe and effective in reducing the symptoms of spasticity and tremor in patients with secondary-progressive or primary progressive multiple sclerosis.

DETAILED DESCRIPTION:
The treatment of MS is far from satisfactory. For acute attacks, high dose corticosteroids seem to reduce the duration of attacks and to reduce the likelihood of future attacks. Immunomodulatory agents, available in this disease over the last decade, reduce the frequency of severe attacks by about one third. The remainder of the treatments are symptomatic, aimed at reducing the disability already present.

Recent research into the CB1 and CB2 cannabinoid receptor systems suggest that cannabis may have the potential for affecting both the pathogenic mechanisms and the symptoms of MS. In light of the autoimmune hypothesis of the etiology of MS, THC could directly alter immune function in a manner that might reduce (or increase) the primary pathology of the disease.

Comparisons: Three treatment arms will be compared: 1) inhaled cannabis and oral placebo, 2) inhaled placebo and oral THC, 3) inhaled placebo and oral placebo, with the effects of these agents analyzed at thirty and sixty days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinically definite multiple sclerosis as defined by Poser criteria
* Primary or secondary disease course
* Moderate or severe spasticity
* Age 21 or older

Exclusion Criteria:

* Preexisting pulmonary conditions, including poorly controlled asthma, chronic bronchitis, emphysema, bronchiectasis, and other significant pulmonary disorders
* Preexisting cardiac conditions, including ischemic heart disease, congestive heart failure, and other significant cardiac disorders
* Inability to abstain from tobacco or marijuana smoking, or use of alcohol or sedative or hypnotic medications during the duration of the study
* Past history of abuse of recreational drugs, including marijuana and alcohol in the last 12 months
* History of or currently meets DSM-IV criteria for dependence on cannabis
* Use of cannabis, marijuana, or THC in the last two weeks
* Preexisting dementia, mania, depression, or schizophrenia or other poorly controlled psychiatric illness
* Exacerbation of MS within 30 days prior to screenin visit
* Current use of cyclophosphamide, mitoxanthrone, or cladribine
* Arthritis, bony and soft tissue disorders interfering with spasticity measures
* Inability to provide informed consent
* Recent cannabis use of more than twice per week one month prior to study entry

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-03; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Change in an objective measurement of spasticity between the pretreatment assessment and the 4- and 8-week assessments.

SECONDARY OUTCOMES:
Differences between active agent and placebo in the changes in Ashworth Scale, Functional System Score, Expanded Disability Status Score, Ambulation Index, Functional Composite Score, and Quality of Life Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Agius, M.D., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

REFERENCES:
- See also: Center for Medicinal Cannabis Research — http://cmcr.ucsd.edu